CLINICAL TRIAL: NCT01509898
Title: The Use of Water Jet for Initial Treatment FOR Peri-Implant Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0374-11-RMB
Record Dates: First submitted 2012-01-01; First posted 2012-01-13 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- water-Jet (Experimental): use of water jet for 1 month
  Interventions: Device: Water jet

INTERVENTIONS:
Device: Water jet — use of water jet for a month
  Other Names: silonit water jet

SUMMARY:
The aim of this study was to evaluate the effect of a dental water jet on initial peri-implant disease resolution.

DETAILED DESCRIPTION:
Peri-implant disease is becoming more frequent during the last decade. Till today, there is no effective evidence-based treatment. The use of water-jet might improve those situations and reduce morbidity and implant loss.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Informed Consent Form.
* Patient suffer from peri- implant disease
* Age Eligible for study: 18 year old and older
* Genders Eligible for study: Both

Exclusion Criteria:

* Patient substantially fails to comply with the study schedule, or treatment program as described in this Protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07-18 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Probing depth | one month
  Probing depth around the implant

SECONDARY OUTCOMES:
Bleeding on probing | one month
  Bleeding on probing (BOP) around the implant

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Liran Levin, DMD, Study Director — Department of periodontology
Locations (1):
- Rambam Hospital, Haifa, Israel